CLINICAL TRIAL: NCT04512742
Title: A Clinical Study to Develop a Controlled Human Infection Model Using Leishmania Major-infected Sand Flies
Acronym: LEISHChallenge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of York (Other)
Collaborators: Medical Research Council (Other Government); Department for International Development, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Paul Kaye, Professor of Immunology, University of York
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LEISH_Challenge
Record Dates: First submitted 2020-08-11; First posted 2020-08-13 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Leishmaniasis; Cutaneous Leishmaniases; Insect Bites
Keywords: Leishmaniasis; Cutaneous Leishmaniases; Controlled Human Infection Model; Human Challenge; Sand Fly; Phlebotomus
MeSH Terms: conditions — Leishmaniasis; Leishmaniasis, Cutaneous; Insect Bites and Stings

STUDY DESIGN:
Intervention Model Description: Controlled human infection study, with an adaptive design. The first six subjects will be exposed to biting by Phlebotomus duboscqi infected by Leishmania major and assess the 'take rate', that is the number of subjects developing parasitologically confirmed cutaneous leishmaniasis (PCCL) lesions. If 6/6 subjects develop PCCL lesions no further recruitment will take place; if only < 6 subjects develop PCCL lesions, then an adaptive design will be followed as described elsewhere.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Leishmania infected-Phlebotomus duboscqi human challenge (Other): There is no clear indication in the medical literature to determine which of the major sand fly vectors of Leishmania major - Phlebotomus papatasi or Phlebotomus duboscqi, will be most effective at transmitting infection to a human host. Both species have a similar mode of feeding and can support L. major development. In our previous study, FLYBITE, no significant difference in biting rates on humans was observed. Based on pre-clinical data , Phlebotomus duboscqi was determined to be the lead candidate for use in this study. If all the 6 participants have developed lesions within the 6-month follow up after Leishmania challenge, the challenge phase of the study is completed. If only 5 participants have developed lesions, then a further 6 participants will undergo Leishmania challenge by P. duboscqi. If only 4 or less subjects in the first cohort develop lesions, then the investigators will switch vector to P. papatasi and a further 6 subjects will undergo Leishmania challenge.
  Interventions: Other: biting by Phlebotomus duboscqi infected with Leishmania major

INTERVENTIONS:
Other: biting by Phlebotomus duboscqi infected with Leishmania major — The first six subjects will be exposed to biting by Phlebotomus duboscqi infected by Leishmania major and assess the 'take rate', that is the number of subjects developing parasitologically confirmed cutaneous leishmaniasis (PCCL) lesions. If 6/6 subjects develop PCCL lesions no further recruitment will take place; if only < 6 subjects develop PCCL lesions, then an adaptive design will be followed.

SUMMARY:
The disease leishmaniasis mainly occurs in hot and tropical countries, affects millions of people and causes around 20,000 deaths across the world every year. Leishmaniasis is caused by the Leishmania parasite and is transmitted by sand flies. The parasite is tiny and not visible to the naked eye, whereas the sand fly is visible but small and inconspicuous.

There are different types of leishmaniasis which can affect the skin (cutaneous leishmaniasis) or the internal organs of the body (visceral leishmaniasis). Some of the milder forms will produce skin problems which will be localised, whilst other forms of leishmaniasis will cause widespread skin changes. The skin lesions of cutaneous leishmaniasis can be disfiguring if left untreated.

There are some treatments for leishmaniasis but many of them are not easy to use or don't work well. Therefore, new treatments are needed including vaccines that prevent or work against leishmaniasis.

A solution being adopted for other diseases, which the investigators now wish to adopt for leishmaniasis is to develop a 'Controlled human infection model' (CHIM). These models involve deliberate exposure of individuals to an infection, in order to better understand how the disease works and to test potential vaccines and treatments. They have contributed knowledge that has led to advances in the development of treatments.

This is study builds on an our initial successful study, FLYBITE, where uninfected (disease-free) sand flies were used to test the safety aspects and ensure that sand flies were able to bite human participants in a controlled environment. The investigators observed no major adverse effects and it was well tolerated by participants. The investigators therefore wish to proceed to a study using sand flies infected with a form of leishmaniasis that causes localised skin disease and is treatable, on the pathway to assessing future vaccines.

DETAILED DESCRIPTION:
This is a clinical study in up to twelve healthy Leishmania-naïve subjects aged between 18 and 50 years old who develop a confirmed sand fly bite. Initially six subjects will be studied and exposed to biting by Phlebotomus duboscqi infected by Leishmania major. An adaptive design will be used, that has been pragmatically designed to minimise unnecessary exposure of volunteers to Leishmania and maximise the likelihood of developing a reproducible Controlled Human Infection Model.

The primary objective is the development of a controlled human infection model of Leishmania major using sand fly transmission which is (a) effective and (b) safe.

The first six subjects will be exposed to biting by Phlebotomus duboscqi (sand fly species) infected by Leishmania major (species of leishmaniasis causing cutaneous, ie skin disease) and assess the 'take rate', that is the number of subjects developing parasitologically confirmed cutaneous leishmaniasis (PCCL) lesions. If 6/6 subjects develop PCCL lesions no further recruitment will take place; if only < 6 subjects develop PCCL lesions, then an adaptive design will be followed.

This study is based on an initial study, entitled FLYBITE (clinicaltrials.gov identifier: NCT03999970).

the FLYBITE study was a clinical study to develop a sand fly biting protocol using pathogen-free blood-fed sand flies. Twelve healthy participants were enrolled into the study and all 12 participants experienced at least one successful sand fly bite.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 50 years on the day of screening
* Willing to give consent for exposure to Leishmania-infected sand fly with the intention of causing a cutaneous leishmaniasis lesion
* Willing and able to give written informed consent
* Willing to undergo Hepatitis B, Hepatitis C & HIV testing
* Willing to undergo a pregnancy test during screening and follow-up visits and must not be breastfeeding
* Willing to refrain from blood donation during the study
* Using a reliable and effective form of contraception (pre-menopausal female participants)
* Judged, in the opinion of a medically qualified Clinical Investigator, to be able and likely to comply with all study requirements as set out in the protocol
* Without any other significant health problems as determined by medical history, physical examination, results of screening tests and the clinical judgment of a medically qualified Clinical Investigator
* Available for the duration of the study
* Willing to refrain from travel to regions where Leishmania-transmitting sand flies are present, from recruitment until an appropriate point (judged by study investigators).
* Willing to consent to a copy of the past medical history to be provided by the participants GP (General Practitioner) practice.
* Agree to registration on a national database of study & trial subjects to prevent over-volunteering (TOPS)
* Willing to give consent for study investigators to contact the participants GP in the event of a significant abnormality being observed
* Willing to show identification documents to confirm identity
* Willing to give consent to biopsy(s) of suspected cutaneous leishmaniasis lesions

Exclusion Criteria:

* Receipt of any vaccine within 21 days of screening
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned study.
* History of significant allergic disease/atopy (e.g. eczema, hay fever, asthma) or reactions; or a history of severe or multiple allergies to drugs or pharmaceutical agents, as judged by the clinical investigators
* Any significant chronic skin condition as judged by the clinical investigators
* Any history of confirmed Leishmaniasis infection
* Any history of travel within the last 30 days to regions where Leishmania major-transmitting sand flies are endemic*.
* Any history of more than 30 continuous days stay in regions where Leishmania major-transmitting sand flies are endemic within the last 10 years*.
* Any history of severe local or general reaction to insect bites, defined as
* Local: extensive, indurated redness and swelling involving most of the antero-lateral thigh or the major circumference of the arm, not resolving within 72 hours
* General: fever ≥ 39.5°C, anaphylaxis, bronchospasm, laryngeal oedema, collapse, convulsions or encephalopathy within 48 hours
* Any history of anaphylaxis
* Females - current pregnancy, less than 12 weeks postpartum, lactating or willingness/intention to become pregnant during the study.
* Any clinically significant abnormal finding on screening biochemistry or haematology blood tests as judged by study investigators
* Total IgE (immunoglobulin E) levels > 214 IU/ml
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months
* A diagnosis of diabetes type 1 or type 2 or significantly raised HbA1c (>48mmol/mol)
* Active Tuberculosis, leprosy, or malnutrition
* Any significant chronic illness requiring hospital specialist input as judged by study investigators
* Any significant psychiatric conditions as judged by general practitioner and/or study clinical team
* Unlikely to comply with the study protocol
* Participating in significant current or recent research (involving an investigational medicinal product or other significant intervention) within the past 3 months (as judged by study investigators)
* Any other significant disease, disorder, finding or medical history, which, in the opinion of a medically qualified Clinical Investigator, may either put the participant at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-10-16 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
The take rate of parasitologically confirmed cutaneous leishmaniasis lesions in study subjects | 1 year
  As the purpose is to develop a Controlled Human Infection Model with a high take rate, and as curative interventions will be carried out very early in the disease course, the P. duboscqi sand fly infected by Leishmania major has been chosen for the first six eligible and consented volunteers.
  The investigators will assess the 'take rate', that is the number of subjects developing parasitologically confirmed cutaneous leishmaniasis (PCCL) lesions. If 6/6 subjects develop PCCL lesions no further recruitment will take place; if only < 6 subjects develop PCCL lesions, then the investigators will follow an adaptive design.
Determine rate of adverse events, determined by data collection through history, clinical examination & blood tests. | 1 year
  The development of any study-associated serious adverse events or grade 3 adverse events at day 3 post-biting will result in a temporary halt and review of the sand fly biting schedule. Therefore the investigators will review the safety outcomes 3 days after all biting procedures in real time for each pair of subjects.
  Successful treatment of cutaneous leishmaniasis lesions in participants, and absence of lesions at 1 year follow up.

SECONDARY OUTCOMES:
Determine rate of cutaneous leishmaniasis lesion development following infected sand fly bite | 1 year
  As determined by clinical examination, then biopsy and parasitological confirmation
Determine response to Leishmania major-infected sand fly bite in terms of immunohistology and immunopathology | 1 year
  Analysis of immune and inflammatory response (for example macrophage and T cell phenotype) and histology compatible with CL.
Determine parasite load in cutaneous leishmaniasis lesions in comparison to number of sand fly bites received and rate of lesion development | 1 year
  By polymerase chain reaction (PCR) analysis of biopsy tissue of lesion site
Determine acceptance and psychological impact of Leishmania major-infected sand fly challenge | 1 year
  Using psychometric questionnaires and focus groups

OTHER OUTCOMES:
Exploratory objectives | 1 year
  In the case of a ≤66% take rate of Leishmania major with Phlebotomus duboscqi, to evaluate the take rate using Phlebotomus papatasi.
  To deep phenotype and compare CL and normal skin biopsies, in those who agree to donate such, using digital spatial profiling of host and parasite mRNA and protein expression, and mass spectroscopy imaging.
  To determine human reactogenicity to Leishmania major-infected sand fly bite in macroscopic, dermoscopic, immunological and biochemical terms

CONTACTS AND LOCATIONS:
Overall Officials: Charles Lacey, BMBS, MD, Principal Investigator — University of York
Locations (1):
- Translational Research Facility, Department of Biology, University of York, York, North Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parkash V, Ashwin H, Dey S, Sadlova J, Vojtkova B, Van Bocxlaer K, Wiggins R, Thompson D, Dey NS, Jaffe CL, Schwartz E, Volf P, Lacey CJN, Layton AM, Kaye PM. Safety and reactogenicity of a controlled human infection model of sand fly-transmitted cutaneous leishmaniasis. Nat Med. 2024 Nov;30(11):3150-3162. doi: 10.1038/s41591-024-03146-9. Epub 2024 Aug 2. PMID 39095597
- [Derived] Parkash V, Jones G, Martin N, Steigmann M, Greensted E, Kaye P, Layton AM, Lacey CJ. Assessing public perception of a sand fly biting study on the pathway to a controlled human infection model for cutaneous leishmaniasis. Res Involv Engagem. 2021 May 30;7(1):33. doi: 10.1186/s40900-021-00277-y. PMID 34053461